CLINICAL TRIAL: NCT05073224
Title: Neuromuscular Biomechanics of the Lumbopelvic Stabilizing Muscles in Nulligravid and Postpartum Women
Brief Title: Muscle Function After Childbirth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carroll University (Other)
Responsible Party: Principal Investigator, Rita Deering, Associate Professor, Carroll University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-0275; A536130 (Other: UW Madison); Protocol Version 6/9/2020 (Other: UW Madison)
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Postpartum; Muscle Fatigue; Force Steadiness; Nulligravid; Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postpartum (Experimental): Participants who are six months postpartum will complete 2 experimental sessions, separated by 7-10 days. Participants will complete multiple questionnaires, maximal voluntary contractions of the lower extremity muscles, clinical tests of lumbopelvic neuromuscular control/posterior pelvic pain provocation, and fatiguing lower extremity/trunk muscle exercise. Ultrasound imaging will be performed to measure inter-recti distance. Wireless Electromyography (EMG) sensors will be used to record EMG and limb steadiness (via Inertial Measurement Units (IMU). Physical activity will be measured by questionnaire and accelerometer.
  Interventions: Diagnostic Test: Active Straight Leg Raise Test; Other: Active Straight Leg Raise Fatigue Task; Other: Lower Extremity Strength Testing; Diagnostic Test: Ultrasound imaging of abdominal wall
- Nulligravid (Active Comparator): Participants who have never been pregnant will complete 2 experimental sessions, separated by 7-10 days. Participants will complete multiple questionnaires, maximal voluntary contractions of the lower extremity muscles, clinical tests of lumbopelvic neuromuscular control/posterior pelvic pain provocation, and fatiguing lower extremity/trunk muscle exercise. Ultrasound imaging will be performed to measure inter-recti distance. Wireless EMG sensors will be used to record EMG and limb steadiness (via IMUs). Physical activity will be measured by questionnaire and accelerometer.
  Interventions: Diagnostic Test: Active Straight Leg Raise Test; Other: Active Straight Leg Raise Fatigue Task; Other: Lower Extremity Strength Testing; Diagnostic Test: Ultrasound imaging of abdominal wall

INTERVENTIONS:
Diagnostic Test: Active Straight Leg Raise Test — The ASLR test is a well-established clinical test that assesses stability of the lumbar spine/pelvis, posterior pelvic pain severity, and ability to activate the abdominal muscles. It is performed in supine. Participants are instructed to raise one leg, with the knee straight, to a heel height of 20 cm. The leg is held at the top for 5 seconds, then slowly lowered to the ground. The participant is asked to report perceived difficulty to raise the leg on a 0 to 5 scale (0=not at all difficult; 5=unable to lift leg) and pain on a 0 to 10 scale (0=no pain; 10=worst possible pain). If difficulty or pain are rated at a 1 or higher, the test is repeated with the researcher providing external compression of the pelvis. If perceived difficulty or reported pain are lower with compression, the test is considered positive for lumbopelvic instability. The test is then repeated on the opposite limb.
  Other Names: ASLR Test
Other: Active Straight Leg Raise Fatigue Task — The protocol is similar to the ASLR test, except that the participant is instructed to maintain the elevated leg off the ground for as long as possible. A biofeedback air cuff will be placed under the participant's lumbopelvic region to assess movement of the spine/pelvis. The cuff will be inflated to 40 mm Hg, and the participant instructed to keep the needle as close to 40 mm Hg as possible throughout the test; no information will be provided on how to affect cuff pressure, but visual feedback of cuff pressure will be provided throughout the task. Ratings of perceived exertion (RPE) and pain will be obtained from participants every 30-60 seconds. Task failure will be defined as a heel height ≤10 cm or a change in cuff pressure ≥20 mm Hg. Both limbs will be tested, but in different sessions. The order of limb testing (dominant vs non-dominant) will be randomized and counter-balanced. Limb dominance will be self-reported.
  Other Names: ASLR Fatigue Task
Other: Lower Extremity Strength Testing — A straight leg raise maximal voluntary contraction (MVC) of each lower extremity an MVC of the hip extensors of the grounded limb will be performed in supine before and within 2 minutes of completing the ASLR fatigue task. The straight leg raise MVC will be performed with a custom-made load cell instrumented strength testing device, which consists of a rigid platform on which the participant will lie. At the foot of the device is a tower that houses 2 load cells connected to a lightly padded push plate.
  The hip extension MVC will be performed on a force plate. Before the ASLR fatigue task, a minimum of 3 MVC trials will be performed for each muscle group, with a minimum of 1 minute rest between trials; the highest peak force will be considered the MVC. Only 1 MVC trial per muscle group will be performed following the ASLR Fatigue Task.
Diagnostic Test: Ultrasound imaging of abdominal wall — Real time ultrasound will be used to assess inter-recti distance above and below the umbilicus. Participants will be assessed with B Mode images in supine at rest, in supine while lifting their head, and in supine while performing a straight leg raise. The Principle Investigator has training and experience in musculoskeletal ultrasound.

SUMMARY:
This study will evaluate lower extremity and trunk neuromuscular control in 78 nulligravid and postpartum women. Participants will attend two experimental sessions, approximately 1 week apart, to assess neuromuscular function. Physical activity levels will also be assessed.

DETAILED DESCRIPTION:
Stability of the lumbar spine and pelvis is essential to nearly all activities of daily living, and is achieved primarily by muscular stabilization. Recent studies have shown that postpartum women are more fatigable than nulligravid women during fatiguing tasks with the lumbopelvic stabilizing muscles (23%) and the trunk flexor muscles (52%) at six months postpartum. Postpartum women also demonstrate impaired control of force with the trunk flexor muscles; however, it is unknown if force control during a fatiguing task of the lumbopelvic stabilizing muscles is impaired in postpartum women.

This study has 3 purposes: (1) To quantify limb steadiness during fatiguing exercise of the lumbopelvic stabilizing muscles among nulligravid women and postpartum women; (2) to quantify muscle activity in the trunk, test limb and contralateral limb to provide insight into motor control; and (3) to identify possible factors (inter-recti distance (IRD), physical activity, pain, biopsychosocial factors) that contribute to neuromuscular function (fatigability and force control).

This is a novel, translational study that, for the first time, will quantify lower extremity force control in postpartum women. As this has not been studied before, to the best of the investigators' knowledge, this proposal will be a pilot study to establish means to utilize in power analyses for future studies of larger magnitude. Furthermore, neuromuscular function is not typically assessed clinically in postpartum women, and no tests exist to easily assess fatigability of the lumbopelvic stabilizing muscles in clinic settings. This study will also provide further data to highlight the ASLR Fatigue Task as a possible clinical examination tool and outcome measure to assess fatigability of the lumbopelvic stabilizing muscles.

ELIGIBILITY:
Inclusion Criteria:

* Post-partum
* Primiparous (this is their first child)

Exclusion Criteria:

* multiple gestation
* prescription anti-inflammatory/pain medications that are taken daily
* significant orthopedic conditions that would contraindicate performance of the fatigue task (such as fractures, severe scoliosis, etc)
* cardiovascular & pulmonary disease
* neuromuscular health conditions (such as diabetes, neuropathy, multiple sclerosis, stroke, seizures, etc)
* history of previous abdominal surgery (with the exception of Cesarean delivery)

Nulligravid Women (Controls)

* Women from the surrounding community will also be recruited to serve as controls
* Nulligravid women will meet the same inclusion/exclusion criteria as the postpartum women, with the exception of never having been pregnant

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Posterior Pelvic Pain | up to 10 days
  The Active Straight Leg Raise (ASLR) test is a well-established clinical test that assesses stability of the lumbar spine/pelvis, posterior pelvic pain severity, and ability to activate the abdominal muscles. It is performed in supine. Participants are instructed to raise one leg, with the knee straight, to a heel height of 20 cm. The leg is held at the top for 5 seconds, then slowly lowered to the ground. The participant is asked to report pain on a 0 to 10 scale (0=no pain; 10=worst possible pain). The test is then repeated on the opposite limb.
Incidence of Perceived Difficulty with ASLR Task | up to 10 days
  The Active Straight Leg Raise (ASLR) test is a well-established clinical test that assesses stability of the lumbar spine/pelvis, posterior pelvic pain severity, and ability to activate the abdominal muscles. It is performed in supine. Participants are instructed to raise one leg, with the knee straight, to a heel height of 20 cm. The leg is held at the top for 5 seconds, then slowly lowered to the ground. The participant is asked to report perceived difficulty to raise the leg on a 0 to 5 scale (0=not at all difficult; 5=unable to lift leg). The test is then repeated on the opposite limb.
Incidence of Lumbopelvic Instability | up to 10 days
  The Active Straight Leg Raise (ASLR) test is a well-established clinical test that assesses stability of the lumbar spine/pelvis, posterior pelvic pain severity, and ability to activate the abdominal muscles. It is performed in supine. Participants are instructed to raise one leg, with the knee straight, to a heel height of 20 cm. The leg is held at the top for 5 seconds, then slowly lowered to the ground. The participant is asked to report perceived difficulty to raise the leg on a 0 to 5 scale (0=not at all difficult; 5=unable to lift leg) and pain on a 0 to 10 scale (0=no pain; 10=worst possible pain). If difficulty or pain are rated at a 1 or higher, the test is repeated with the researcher providing external compression of the pelvis. If perceived difficulty or reported pain are lower with compression, the test is considered positive for lumbopelvic instability. The test is then repeated on the opposite limb.
Mean Time to ASLR Fatigue Task Failure | up to 10 days
  For the ASLR Fatigue Task, the participant is instructed to maintain the elevated leg off the ground for as long as possible. Task failure will be defined as a heel height greater than or equal to 10 centimeters off the ground.
Maximum Lower Extremity Strength: Leg | up to 10 days
  A straight leg raise maximal voluntary contraction (MVC) of each lower extremity will be performed in the supine position before and within 2 minutes of completing the ASLR fatigue task with a custom made load cell instrumented strength testing device. This device consists of a rigid platform on which the study participant will lie supine. At the foot of the device is a tower that houses 2 load cells and is connected to a lightly padded push plate. This push plate can be raised and lowered such that the participant can push up into the plate (contacts the anterior surface of the participant's shin) or push down onto the push plate (contacts the posterior aspect of the participant's heel).
  Before the ASLR fatigue task, a minimum of 3 MVC trials will be performed on each leg, with a minimum of 1 minute rest between trials, in order to ensure a true maximum has been obtained; the highest peak force will be considered the MVC. Only 1 MVC trial per leg will be performed following the
Maximum Lower Extremity Strength: Hip Extension | up to 10 days
  A hip extension MVC will also be performed in supine (pushing down into the ground) on a force plate (1000 Hz) prior to performance of the ASLR fatigue task. Only the leg that will remain in contact with the force plate during the ASLR fatigue task (grounded limb) will perform the extension MVC, in order to normalize downward pressure into the force plate by the grounded limb during performance of the ASLR fatigue task. This will allow us to quantify activity of the grounded limb during the fatiguing task. A minimum of 3 hip extension MVCs will be performed, with 1 minute rest between trials. An MVC may also be assessed at the end of the fatiguing exercise bout.
Limb Steadiness Measured by Limb Acceleration | up to 10 days
  An inertial measurement unit (Trigno, Delsys, Boston, MA) will be placed on the test limb to track movement of the limb during performance of the ASLR Fatigue Task. Fluctuations in limb acceleration will be measured and quantified as the standard deviation of acceleration. Limb steadiness will be collected online, stored, and analyzed offline with ConsensysPRO software. The investigators hypothesize that fluctuations in limb acceleration will be greater among postpartum women as compared to nulligravid women during the performance of the ASLR Fatigue Task.
Abdominal Fascial Integrity Measured by Mean Inter-Recti Distance | up to 10 days
  Real time ultrasound will be used to assess inter-recti distance above and below the umbilicus. Participants will be assessed with B Mode images in supine at rest, in supine while lifting their head, and in supine while performing a straight leg raise.

SECONDARY OUTCOMES:
Assessment of fatigability of the lumbopelvic stabilizing muscles measured by the ASLR Fatigue Task: Mean Ratings of Perceived Exertion (RPE) | up to 10 days
  For the ASLR Fatigue Task, the participant is instructed to maintain the elevated leg off the ground for as long as possible. A biofeedback air cuff placed under the participant's lumbopelvic region assesses movement of the spine/pelvis during the test. The cuff will be inflated to 40 mm Hg, and the participant will be instructed to keep the needle as close to 40 mm Hg as possible throughout the test. Ratings of perceived exertion (RPE, from 0-10 with higher scores increased exertion) are measured every 30-60 seconds. Task failure will be defined as a heel height ≤10 cm or a change in cuff pressure ≥20 mm Hg. Both limbs will be tested in different sessions.
Assessment of fatigability of the lumbopelvic stabilizing muscles measured by the ASLR Fatigue Task: Mean Pain Score | up to 10 days
  For the ASLR Fatigue Task, the participant is instructed to maintain the elevated leg off the ground for as long as possible. A biofeedback air cuff placed under the participant's lumbopelvic region assesses movement of the spine/pelvis during the test. The cuff will be inflated to 40 mm Hg, and the participant will be instructed to keep the needle as close to 40 mm Hg as possible throughout the test. Pain Scores will be measured (0-10 with higher scores increased pan) every 30-60 seconds. Task failure will be defined as a heel height ≤10 cm or a change in cuff pressure ≥20 mm Hg. Both limbs will be tested in different sessions.
Average Total Activity Counts (TAC) per day over 7 days | up to 7 days
  Physical activity habits around the time of testing will be assessed with a tri-axial accelerometer for 7 days outside of the laboratory, in part by measuring the TAC per day. TAC is the total number of filtered, full-wave rectified, integrated accelerations (all directions). These will then be averaged/day based on the total number of valid wear days for each participant.
Physical Activity Measured by Average Steps per day over 7 days | up to 7 days
  Physical activity habits around the time of testing will be assessed with a tri-axial accelerometer for 7 days outside of the laboratory, in part by measuring mean steps per day.
  This will be quantified as reported by the ActiGraph accelerometer and ActiLife analysis software, which uses the vertical axis data. The Algorithm used by ActiGraph is not publicly available, but ActiGraph accelerometers are frequently used in research quantifying physical activity.
Mean Duration per day of Moderate-Vigorous Physical Activity (MVPA) over 7 days: tri-axial counts | up to 7 days
  Physical activity habits around the time of testing will be assessed with a tri-axial accelerometer for 7 days outside of the laboratory, in part by measuring mean duration per day of MVPA.
  Intensity of physical activity assessed using tri-axial counts (per the accelerometer software) are as follows: Light physical activity is between 200 and 2690 counts/min, moderate intensity between 2690-6166 counts/min, and vigorous intensity is ≥ 6167 counts/min. MVPA is ≥2690.
Mean Duration per day of Moderate-Vigorous Physical Activity (MVPA) over 7 days: vertical counts | up to 7 days
  Physical activity habits around the time of testing will be assessed with a tri-axial accelerometer for 7 days outside of the laboratory, in part by measuring mean duration per day of MVPA.
  Intensity of physical activity assessed using vertical counts (per the accelerometer software) are as follows: Light physical activity is between 100 and 759 counts/min, moderate intensity is 760-5999 counts/min, and vigorous intensity is ≥ 6000 counts/min (MVPA is > 760 counts/min).
Average Minutes per Day of Activity in at least 5-minute bouts | up to 7 days
  Physical activity habits around the time of testing will be assessed with a tri-axial accelerometer for 7 days outside of the laboratory, in part by measuring mean duration per day of all activity.
  Average minutes per day of activity within each of the following categories: light = 25.8 mg - 100.5 mg; moderate = 100.6 mg - 428.7 mg; vigorous = > 428.8 mg
  (mg is the vector magnitude of acceleration calculated in gravities using Euclidean Norm minus 1 metric)
Average Minutes per Day of Activity in at least 10-minute bouts | up to 7 days
  Physical activity habits around the time of testing will be assessed with a tri-axial accelerometer for 7 days outside of the laboratory, in part by measuring mean duration per day of all activity.
  Average minutes per day of activity within each of the following categories: light = 25.8 mg - 100.5 mg; moderate = 100.6 mg - 428.7 mg; vigorous = > 428.8 mg.
  (mg is the vector magnitude of acceleration calculated in gravities using Euclidean Norm minus 1 metric)
Percent Change in Global Surface EMG Recordings: Abdominal Muscles | up to 10 days
  EMG will be reported as the root mean square (RMS) value. The percent change in EMG from the start of the task to task failure will be examined.
Percent Change in Global Surface EMG Recordings: Rectus femoris | up to 10 days
  EMG for the rectus femoris will be normalized to the maximum RMS EMG obtained during lower extremity strength testing. The percent change in EMG from the start of the task to task failure will be examined.
Mean Global Pittsburgh Sleep Quality Index (PSQI) Score | up to 10 days
  The PSQI assesses seven sleep domains: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. The seven components scores are then added to yield a global PSQI score in the range of zero to 21. Higher scores indicate worse sleep quality. A global score greater than five is diagnostic of poor sleep quality.
Mean Pelvic Floor Distress Inventory Short Form (PFDI-20) Score | up to 10 days
  The PFDI-20 is composed of 20 items total on three scales (Pelvic Organ Prolapse, Colorectal-Anal Distress, Urinary Distress), each scored on a 5 point likert scale. Mean scores from each scale are calculated and multiplied by 25, then added together for a total possible range of scores from 0-300. Higher scores indicate increased pelvic floor distress.
Mean Oswestry Disability Index Score | up to 10 days
  This disability index measures how much lower back or leg pain affects the ability to manage everyday life. There are 10 sections, each section is scored from 0-5 for a total possible range of scores 0-50. The resultant score is divided by the total possible score and multiplied by 100 to get a percentage of disability.
Mean Pain Catastrophizing Scale (PCS) Score | up to 10 days
  The PCS is a measure of thoughts and feelings when one is in pain. It is a 13 item questionnaire scored on a 5 point likert scale. The total possible range of scores is 0-52 where higher scores indicate a higher degree of overwhelm with respect to pain.
Mean Edinburgh Postnatal Depression Scale (EPDS) Score | up to 10 days
  The EPDS is a 10-item survey that screens for symptoms of depression that have been present in the previous 7 days. Each question is scored on a 4-point scale ranging from 0 to 3 points for a total possible range of scores between 0-30, where higher scores indicate increased depression. Only postpartum participants will complete this survey.
Mean Post Traumatic Stress Disorder (PTSD) Score | up to 10 days
  The PTSD Checklist for DSM-5 with Life Events Checklist for DSM-5 and Criterion A scale will be used to assess participant level of PTSD. The measure has a total range of scores between 0-80 with higher scores indicating greater PTSD symptoms.
  Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5)
Mean Tampa Scale for Kinesiophobia (TSK) Score | up to 10 days
  The TSK scale measures fear of movement. The total possible range of scores is 17-68, where higher score means higher degree of kinesiophobia.
Mean Pelvic Girdle Questionnaire (PGQ) Score | up to 10 days
  The PGQ is a measure of how much pelvic girdle pain affects daily activities. It is a 25-item questionnaire scored on a 4 point likert scale for a total possible range of scores from 0-75 where higher scores indicate increased burden on daily activities.

OTHER OUTCOMES:
Root mean square (RMS) of global EMG | up to 10 days
  Muscle behavior will be quantified from surface EMG recordings of the rectus abdominis and rectus femoris using multi-channel array surface EMG electrodes during maximal and submaximal contractions and fatiguing exercise of the abdominal muscles. If successful, RMS of global EMG will be reported.
Percent of Maximum Voluntary Isometric Contraction (MVIC) | up to 10 days
  Muscle activity will be quantified from surface EMG recordings of the rectus abdominis and rectus femoris using a multi-channel array surface EMG electrodes during submaximal contractions and fatiguing exercise of the abdominal muscles, and normalized to the RMS EMG during maximal voluntary isometric contractions (MVIC). If successful, percent of MVIC will be reported.
Mean discharge rate of single motor units | up to 10 days
  Single motor unit behavior will be extracted from surface EMG recordings of the rectus abdominis and rectus femoris using a multi-channel array surface EMG electrodes during submaximal contractions and fatiguing exercise of the abdominal muscles, as an exploratory analysis. If successful, mean discharge rate of single motor units will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Deering, PT, DPT, PhD, Principal Investigator — Carroll University
Locations (1):
- Carroll University, Waukesha, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No